CLINICAL TRIAL: NCT01006252
Title: A Randomized Phase 3 Study of Tasisulam-sodium Administered as an Intravenous Infusion on Day 1 of a 28-Day Cycle Versus Paclitaxel as Second-line Treatment in Patients With Metastatic Melanoma
Brief Title: A Study of Tasisulam-sodium Versus Paclitaxel as Treatment for Metastatic Melanoma
Acronym: SUMMIT-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: More possibly treatment-related deaths on tasisulam-sodium arm.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13101; H8K-MC-JZAO (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Melanoma
Keywords: metastatic; second-line
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tasisulam-sodium (Experimental): Individualized tasisulam-sodium dose was dependent on participant's height, weight, and gender. Dose was adjusted based on laboratory parameters. Treatment was administered intravenously on Day 1 of a 28-day cycle, until disease progression.
  Interventions: Drug: Tasisulam-sodium
- Paclitaxel (Active Comparator): Paclitaxel 80 milligrams per square meter (mg/m^2) administered intravenously on Days 1, 8, and 15 of a 28-day cycle, until disease progression
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Tasisulam-sodium — Administered intravenously on Day 1 of a 28-day cycle, until disease progression.
  Other Names: LY573636
  Arms: Tasisulam-sodium
Drug: Paclitaxel — 80 mg/m^2 administered intravenously on Days 1, 8, and 15 of a 28-day cycle, until disease progression
  Arms: Paclitaxel

SUMMARY:
The primary purpose of this study was to see how tasisulam-sodium affected metastatic melanoma when compared against paclitaxel as measured by overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologic and/or cytologic diagnosis of metastatic melanoma (Stage IV).
* Have the presence of evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.0).
* Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Have progressed after 1 previous systemic treatment containing dacarbazine or temozolomide for metastatic melanoma.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, or other investigational therapy for at least 30 days (6 weeks for mitomycin-C or nitrosoureas) before study enrollment and recovered from the acute effects of therapy (except alopecia).
* Have a serum albumin level greater than or equal to 3.0 grams per deciliter (g/dL) or greater than or equal to 30 grams per liter (g/L).

Exclusion Criteria:

* Have received greater than or equal to 2 previous chemotherapy-containing systemic treatment regimens for metastatic melanoma. An immunotherapy or antibody-based regimen (including biologic agents and vaccination-based treatments), or treatment with a targeted agent (for example, BRAF or c-Kit inhibitor is not counted as a prior treatment regimen for determining study eligibility, unless either was combined with a cytotoxic drug).
* Have active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of study entry. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before study entry to rule out occult brain metastasis. Participants with a history of a solitary CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) and not requiring steroids are eligible.
* Are receiving warfarin.
* Have primary ocular or mucosal melanoma.
* Any previous treatment with paclitaxel or a paclitaxel-containing regimen for metastatic melanoma.
* Have serious concomitant disorders, including active bacterial, fungal, or viral infection, incompatible with the study (at the discretion of the investigator).
* Have previously completed or withdrawn from this study or any other study investigating tasisulam-sodium.
* Have a known hypersensitivity to paclitaxel or Cremophor EL (polyoxyethylated castor oil).
* Are pregnant or lactating.
* Have received a recent (within 30 days before enrollment) or are receiving concurrent yellow fever vaccination.
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb).
* Are unable to withhold dosing of non-steroidal anti-inflammatory drugs (NSAIDs) or proton-pump inhibitors (PPIs) for at least 72 hours before and after treatment with tasisulam-sodium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (122):
- United States (50):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakeland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Park Ridge, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goshen, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westwood, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morristown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Porte, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coffs Harbour, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Townsville, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif
- Germany (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buxtehude
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heilbronn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quedlinburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- Norway (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oslo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trondheim
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otwock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
- United Kingdom (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hampstead, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northwood, Middlesex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel: Paclitaxel 80 mg/m^2 administered intravenously on Days 1, 8, and 15 of a 28-day cycle, until disease progression
Period: Overall Study
Arm/Group | Tasisulam-sodium | Paclitaxel
Started | 168 | 168
Received Treatment | 164 | 161
Completed | 168 | 168
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasisulam-sodium | Paclitaxel | Total
Number analyzed (Participants) | 168 | 168 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.30 (13.20) | 59.44 (13.43) | 58.87 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 103 | 105 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 84 | 75 | 159
  Unknown or Not Reported | 83 | 89 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 158 | 162 | 320
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 50 | 90
  Finland | 1 | 2 | 3
  Spain | 3 | 7 | 10
  Austria | 5 | 3 | 8
  Israel | 3 | 3 | 6
  United Kingdom | 8 | 1 | 9
  Italy | 8 | 11 | 19
  France | 32 | 26 | 58
  Canada | 4 | 8 | 12
  Poland | 7 | 6 | 13
  Belgium | 7 | 6 | 13
  Australia | 1 | 5 | 6
  Norway | 5 | 5 | 10
  Germany | 32 | 28 | 60
  Sweden | 3 | 3 | 6
  South Korea | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is duration from enrollment to death; OS censored for participants who were alive at last contact.
Time Frame: Randomization to date of death from any cause (assessed at every cycle and every 60 days following treatment discontinuation) up to 14.32 months
Population: The intent-to-treat (ITT) analysis population included all participants randomized to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 168 | 168
months | 6.77 [5.88 to 8.28] | 9.36 [6.90 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.121, Stratified log rank — Statistical significance was assessed at an alpha level of 0.05; Hazard Ratio (HR) = 1.23

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is time from date of first dose to first observation of disease progression (PD); PD=20% increase in sum of the longest diameter of target lesions, or death from any cause.
Time Frame: Randomization to date of objectively determined PD, or death from any cause (assessed at every cycle and every 60 days following treatment discontinuation) up to 13.70 months
Population: The intent-to-treat (ITT) analysis population included all participants randomized to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 168 | 168
months | 1.94 [1.87 to 2.04] | 2.14 [1.91 to 2.96]
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.048, Stratified log rank — Statistical significance was assessed at an alpha level of 0.05; Analysis adjusted for Baseline Lactate Dehydrogenase (LDH); Disease Stage; Sex; Previous Single Agent Immunotherapy Treatment; Age Group; Hazard Ratio (HR) = 1.30

3. Secondary Outcome: Percentage of Randomized Participants Having a Confirmed Best Response of Partial Response (PR) or Complete Response (CR)
Description: Response Evaluation Criteria In Solid Tumors (RECIST) criteria: CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; Progressive disease (PD)=20% increase in sum of the longest diameter of target lesions.
Time Frame: First date RECIST criteria met for CR or PR (whichever occurred first) until first date of documented PD, or death from any cause (assessed every other cycle) up to 13.70 months
Population: The intent-to-treat (ITT) analysis population included all participants randomized to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 168 | 168
percentage of participants
  CR | 0 [0 to 0] | 0 [0 to 0]
  PR | 3.0 [0.4 to 5.5] | 4.8 [1.5 to 8.0]
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.396, Unadjusted normal distribution — Statistical significance was assessed at an alpha level of 0.05; Unadjusted normal-distribution approximation for the difference in rates

4. Secondary Outcome: Duration of Response (DoR) for Participants Having an Objective Response of Partial Response (PR) or Complete Response (CR)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; Progressive disease (PD)=20% increase in sum of the longest diameter of target lesions. Analysis was adjusted for Baseline Lactate Dehydrogenase (LDH); Disease Stage; Sex; Previous Single Agent Immunotherapy Treatment; Age Group. Due to limited number of responses for either treatment arm, DoR analysis was not performed.
Time Frame: as for outcome 3
Population: Zero participants analyzed. Duration of Response for CR and PR data was not collected for analysis per study report.
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Randomized Participants Having a Confirmed Best Overall Response of Partial Response (PR) or Complete Response (CR) Plus Participants With an Overall Response of Stable Disease (SD)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; SD=small changes that do not meet above criteria; PD=20% increase in sum of the longest diameter of target lesions.
Time Frame: First date RECIST criteria met for CR, PR, or SD until first date of documented progressive disease (PD), or death from any cause (assessed every other cycle) up to 13.70 months
Population: The intent-to-treat (ITT) analysis population included all participants randomized to treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 168 | 168
percentage of participants | 30.4 [23.4 to 37.3] | 33.9 [26.8 to 41.1]
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.483, Unadjusted normal distribution — Statistical significance was assessed at an alpha level of 0.05; Unadjusted normal-distribution approximation for the difference in rates

6. Secondary Outcome: Time to Deterioration in the Functional Assessment of Cancer Therapy-Melanoma Trial Outcome Index (FACT-M TOI) Score
Description: FACT-M measures domains of health-related quality of life (HR-QoL): physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns of melanoma. FACT-M TOI is the sum of FACT-M physical well-being, functional well-being, and melanoma subscales. Scores range from 0 to 120; Higher scores=better quality of life (QoL). FACT-M TOI score deterioration was defined as time from randomization to a minimally important difference in TOI score or death.
Time Frame: Randomization to first date of deterioration in FACT-M TOI, or death from any cause (assessed every cycle and up to 30 days following treatment discontinuation) up to 13.21 months
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 136 | 141
months | 2.96 [2.30 to 3.71] | 3.52 [2.99 to 4.01]
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.505, Stratified log rank — Statistical significance was assessed at an alpha level of 0.05; Hazard Ratio (HR) = 1.11

7. Secondary Outcome: Change From Baseline at Cycle 2 in Functional Assessment of Cancer Therapy-Melanoma (FACT-M) up to 30 Days Following Treatment Discontinuation
Description: FACT-M measures domains of health-related quality of life (HR-QoL): physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns of melanoma. Total scores range from 0 to 172; Higher scores=better HR-QoL. Least Squares (LS) Mean value was adjusted for treatment group, cycle, treatment-by-cycle interaction, age, Eastern Cooperative Oncology Group (ECOG) performance status, stage of disease at study entry, and best response to previous chemotherapy.
Time Frame: Baseline at Cycle 2, up to 30 days following treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 136 | 141
units on a scale | -0.81 (2.38) | -1.07 (2.40)
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.902, Mixed Model Repeated Measures (MMRM) — P-value given for Overall Main Treatment Effect from the repeated measure model where time was a class variable. Statistical significance was assessed at an alpha level of 0.05; MMRM analyses limited to first 4 cycles due to sparse data; data from 30-day follow-up visit coded to first cycle after last on-treatment cycle
Statistical Analysis 2: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.970, Mixed Model Repeated Measures (MMRM) — P-value given for Treatment-By-Cycle Interaction from the repeated measure model where time was a class variable. Statistical significance was assessed at an alpha level of 0.05; [statistical method as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline at Cycle 3 in Functional Assessment of Cancer Therapy-Melanoma (FACT-M) up to 30 Days Following Treatment Discontinuation
Description: as for outcome 7
Time Frame: Baseline at Cycle 3, up to 30 days following treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Tasisulam-sodium: Individualized tasisulam-sodium dose was dependent on participant's height, weight, and gender. Dose was adjusted based on laboratory parameters. Treatment was administered intravenously on Day 1 of a 28-day cycle until disease progression.
- Paclitaxel: Paclitaxel 80 mg/m^2 administered intravenously on Days 1, 8, and 15 of a 28-day cycle until disease progression.
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 117 | 118
units on a scale | -4.06 (2.47) | -4.69 (2.51)

9. Secondary Outcome: Change From Baseline at Cycle 4 in Functional Assessment of Cancer Therapy-Melanoma (FACT-M) up to 30 Days Following Treatment Discontinuation
Description: as for outcome 7
Time Frame: Baseline at Cycle 4, up to 30 days following treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 46 | 50
units on a scale | -2.86 (2.66) | -2.98 (2.69)
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.902, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 7, analysis 1]; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.970, Mixed Model Repeated Measures (MMRM) — P-value given for Overall Treatment-By-Cycle Interaction from the repeated measure model where time was a class variable. Statistical significance was assessed at an alpha level of 0.05; [statistical method as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline at Cycle 2 in EuroQol-5 Dimensions (EQ-5D) up to 30 Days Following Treatment Discontinuation
Description: EQ-5D consists of 5 items that assess participant's overall health. Participants choose 1 of 3 options that best describe the status of each item. EQ-5D United Kingdom (UK)-based index scores range from -0.59 (worst health) to 1.0 (1.0=perfect health; Positive change from baseline=health improvement). Least Squares (LS) Mean value was adjusted for treatment group, cycle, treatment-by-cycle interaction, age, Eastern Cooperative Oncology Group (ECOG) performance status, stage of disease at study entry, and best response to previous chemotherapy.
Time Frame: Baseline at Cycle 2, up to 30 days following treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 133 | 134
units on a scale | 0.01 (0.03) | -0.00 (0.03)
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.547, Mixed Model Repeated Measures (MMRM) — P-value given for Main Treatment Effect from the repeated measure model where time was a class variable. Statistical significance was assessed at an alpha level of 0.05; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.414, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 7, analysis 2]; [statistical method as in outcome 7, analysis 1]

11. Secondary Outcome: Change From Baseline at Cycle 3 in EuroQol-5 Dimensions (EQ-5D) up to 30 Days Following Treatment Discontinuation
Description: EQ-5D consists of 5 items that assess participant's overall health. Participants choose 1 of 3 options that best describe status of each item. EQ-5D United Kingdom (UK)-based index scores range from -0.59 (worst health) to 1.0 (1.0=perfect health; Positive change from baseline=health improvement). Least Squares (LS) Mean value was adjusted for treatment group, cycle, treatment-by-cycle interaction, age, Eastern Cooperative Oncology Group (ECOG) performance status, stage of disease at study entry, and best response to previous chemotherapy.
Time Frame: Baseline at Cycle 3, up to 30 days following treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 80 | 77
units on a scale | -0.01 (0.03) | -0.06 (0.03)

12. Secondary Outcome: Change From Baseline at Cycle 4 Baseline in EuroQol-5 Dimensions (EQ-5D) up to 30 Days Following Treatment Discontinuation
Description: as for outcome 11
Time Frame: Baseline at Cycle 4, up to 30 days after treatment discontinuation
Population: The analysis population included all randomized participants who had baseline and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasisulam-sodium | Paclitaxel
Number analyzed (Participants) | 42 | 43
units on a scale | -0.05 (0.04) | -0.05 (0.04)
Statistical Analysis 1: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.547, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; [statistical method as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Tasisulam-sodium vs Paclitaxel; Test type: Superiority or Other; p = 0.414, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 7, analysis 2]; [statistical method as in outcome 7, analysis 1]

13. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) During Cycle 1
Time Frame: After drug infusion in Cycle 1 (5 samples drawn over the 28-day cycle)
Population: The analysis population included all participants who received at least 1 dose of study drug for whom PK data were available. PK analysis were only performed on Tasisulam per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- Tasisulam: Dose was adjusted based on participant laboratory parameters and lean body weight; administered intravenously every 28 days until disease progression, or other criteria for participant discontinuation were met.
Arm/Group | Tasisulam
Number analyzed (Participants) | 162
microgram per milliliter (µg/mL) | 375 (14.8)

14. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) During Cycle 2
Time Frame: After drug infusion in Cycle 2 (2 samples drawn over the 28-day cycle)
Population: The analysis population included all participants who received at least 2 doses of study drug for whom pharmacokinetic data were available. PK analysis were only performed on Tasisulam per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Tasisulam
Number analyzed (Participants) | 129
µg/mL | 361 (16.8)

ADVERSE EVENTS:
Description: All randomized participants who received treatment.
Arm/Group | Tasisulam-sodium | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 53/164 | 44/161
Other Adverse Events (participants affected / at risk) | 149/164 | 146/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasisulam-sodium (N=164) | Paclitaxel (N=161)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (19) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Hyperthermia (General disorders) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasisulam-sodium (N=164) | Paclitaxel (N=161)
Anaemia (Blood and lymphatic system disorders) | 15 (17) | 19 (21)
Neutropenia (Blood and lymphatic system disorders) | 13 (17) | 19 (27)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (28) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 4 (4)
Constipation (Gastrointestinal disorders) | 14 (16) | 23 (24)
Diarrhoea (Gastrointestinal disorders) | 31 (39) | 29 (35)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 9 (10)
Nausea (Gastrointestinal disorders) | 29 (33) | 36 (37)
Vomiting (Gastrointestinal disorders) | 16 (17) | 21 (21)
Asthenia (General disorders) | 10 (10) | 19 (21)
Fatigue (General disorders) | 50 (52) | 47 (50)
Oedema peripheral (General disorders) | 12 (14) | 15 (15)
Pyrexia (General disorders) | 17 (18) | 14 (15)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22) | 20 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 13 (14)
Dizziness (Nervous system disorders) | 5 (5) | 10 (11)
Dysgeusia (Nervous system disorders) | 10 (10) | 5 (5)
Headache (Nervous system disorders) | 22 (29) | 12 (13)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 9 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 11 (12)
Insomnia (Psychiatric disorders) | 5 (5) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 21 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 19 (20)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15) | 51 (52)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13) | 9 (11)
Rash (Skin and subcutaneous tissue disorders) | 23 (29) | 23 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days